CLINICAL TRIAL: NCT02626559
Title: Serum Bupivacaine Concentration Levels After Injection of the Knee Joint With a Mixture of Liposomal Bupivacaine and Free Bupivacaine During Total Knee Arthroplasty
Brief Title: Serum Bupivacaine Concentration Levels After Injection of Liposomal Bupivacaine Into the Knee
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Michael Buys, Assistant Professor, University of Utah
Other Study IDs: IRB_00082660
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: liposomal bupivacaine/plain bupivacaine peri-articular injection — Injection of a mixture of liposomal and plain bupivacaine around the knee during total knee arthroplasty.

SUMMARY:
Serum levels of bupivacaine over time after peri-articular injection of a mixture of liposomal bupivacaine and plain bupivacaine during total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Adults of at least 18 years of age having a primary, unilateral total knee arthroplasty with a surgical plan to have an intra-articular injection of a mixture of 266 mg of Exparel, 125 mg of bupivacaine, 1:300,000 epinephrine, and 0.9% saline to make a total volume of 100 ml.

Exclusion Criteria:

* Known hepatic dysfunction or renal insufficiency (creatinine > 1.5 mg/dL);
* allergy to the study medications;
* pregnancy;
* incarceration;
* inability to communicate with the investigators;
* morbid obesity (body mass index > 40 kg/m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults of at least 18 years of age having a primary, unilateral total knee arthroplasty with a surgical plan to have an intra-articular injection of a mixture of 266 mg of Exparel, 125 mg of bupivacaine, 1:300,000 epinephrine, and 0.9% saline to make a total volume of 100 ml.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Serum Bupivacaine levels | 5 minutes to 24 hours after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Uutah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buys MJ, Murphy MF, Warrick CM, Pace NL, Gililland JM, Pelt CE, Bankhead BR, Patzkowsky JL, Johnson KB. Serum Bupivacaine Concentration After Periarticular Injection With a Mixture of Liposomal Bupivacaine and Bupivacaine HCl During Total Knee Arthroplasty. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):582-587. doi: 10.1097/AAP.0000000000000636. PMID 28727583